CLINICAL TRIAL: NCT05808712
Title: Developing Patient-centered Interventions to Improve the Quality of Care in Relationship to Aborted Cancer Surgery
Brief Title: Quality of Care in Relationship to Aborted Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jenny Drott, RN, PhD, Associate Professor, Linkoeping University
Other Study IDs: ACS
Record Dates: First submitted 2023-03-28; First posted 2023-04-11 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Gastrointestinal Cancer
Keywords: cancer nursing,; patient preferences; patient-centered care
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms; Patient Preference | interventions — Validation Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Translation and validation design: To translate the English version of The Supportive Care Needs Survey-short form (SCNS-SF34) questionnaire into Swedish and to test the reliability and validity.
  Design: Translation and validation design
  A multicenter national validation study, in three university hospital in Sweden. Consecutive sampling procedure during a one-year period (2023), to evaluate internal consistency and test-retest reliability of the SCNS-SF34 in Swedish. Number is calculated to be 300 patients, and test-rest (reliability) in 50 patients. Inclusion criteria = >18 years, cancer patients with different gastrointestinal cancer diagnosis. Exclusion criteria= not able to answer a questionnaire in Swedish.
  Demographical and clinical data will be collected using a case report form. The survey will be distributed to patients via a web-based questionnaire or paper and pen questionnaire procedure.
  Interventions: Other: validation

INTERVENTIONS:
Other: validation — Translation and validation design

SUMMARY:
Surgery is often a central curative treatment for gastrointestinal tumors. Surgical treatment of diagnosed cancer tumors is decided after a comprehensive assessment of the patient's physical status, radiological assessments and after careful evaluation at the multidisciplinary conference. Despite the careful preoperative assessment of patients for curative surgery, the planned operation may unexpectedly need to be canceled. Of the patients who were planned for curative resection for pancreatic cancer in 2021 in Sweden, 90% received the intended surgery, and 10% of planned surgery was canceled. The reason for this was disseminated cancer or locally advanced disease in which radical resection is considered impossible to carry out. A systematic review of knowledge reveals a significant lack of evidence regarding patient-centered research and aborted cancer surgery.

The studies in the project have different study designs and methods, and include focus group interviews with staff, translation and validation of a questionnaire to measure care needs, estimation of supportive care needs and patient experiences.

An improved understanding and knowledge of patients' preferences and needs is needed to design interventions that can improve health-related quality of life. This project is dedicated to studying patients undergoing aborted cancer surgery, with the aim of improving the quality of care and meeting patients' care needs.

DETAILED DESCRIPTION:
The overall objective of this research project is to:

* describe the patients experiences and assess supportive care needs following aborted cancer gastrointestinal surgery
* increase knowledge of the healthcare professionals' experiences of aborted cancer surgery from a multi-professional and continuum of cancer care perspective
* increase our clinical knowledge of patient preferences and healthcare professionals' perspective to develop tailored patient-centered interventions with the goal to improve quality of cancer care

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* cancer patients with different gastrointestinal cancer diagnosis

Exclusion Criteria:

- not able to answer the questionnarie SCNS-SF34 in Swedish.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cancer patients with different gastrointestinal cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
supportive care needs, questonnarie | March 2023 - March 2024
  psychometric properties in the swedish version of the questionnarie SCNS-SF34
Rate of supportive care needs in cancer | March 2023 - March 2024
  assessment of supportive care needs via the questionnarie SCNS-SF34 (in Swedish)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Drott, Principal Investigator — Kirurgiska kliniken, Region Östergötland
Locations (2):
- Sweden (2):
  - Jenny Drott, Linköping
  - Department of Surgery, Linköping

IPD SHARING:
Plan to Share IPD: No